CLINICAL TRIAL: NCT01100372
Title: Randomized Phase II AGO-Study Comparing Combined Liposomal Doxorubicin (Myocet) and Gemcitabine (Gemzar) With Liposomal Doxorubicin (Myocet) Monotherapy in Platinum-Refractory and Platinum-Resistant Epithelial Cancer of the Ovary, Fallopian Tube and the Peritoneum
Brief Title: Liposome-Encapsulated Doxorubicin Citrate With or Without Gemcitabine Hydrochloride in Treating Patients With Ovarian Epithelial Cancer, Fallopian Tube Cancer, or Primary Peritoneal Cavity Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University Innsbruck (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000669716; MUI-AGO-10; EUDRACT-2008-008746-20; EU-21028
Record Dates: First submitted 2010-04-07; First posted 2010-04-08 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2010-04

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; recurrent fallopian tube cancer; recurrent primary peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Gemcitabine

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: liposome-encapsulated doxorubicin citrate
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as liposome-encapsulated doxorubicin citrate and gemcitabine hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known whether liposome-encapsulated doxorubicin citrate is more effective when given together with or without gemcitabine hydrochloride in killing tumor cells.

PURPOSE: This randomized phase II trial is studying liposome-encapsulated doxorubicin citrate given together with gemcitabine hydrochloride to see how well it works compared with liposome-encapsulated doxorubicin citrate alone in treating patients with ovarian epithelial cancer, fallopian tube cancer, or primary peritoneal cavity cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the response rate to liposome-encapsulated doxorubicin citrate and gemcitabine hydrochloride versus liposome-encapsulated doxorubicin citrate alone in patients with platinum-refractory or platinum-resistant ovarian epithelial, fallopian tube, or primary peritoneal cavity cancer.

Secondary

* To assess the quality of life of patients treated with these regimens.
* To determine the progression-free and overall survival of patients treated with these regimens.
* To determine the toxicity of these regimens.

OUTLINE: This is a multicenter study. Patients are stratified according to disease (platinum-refractory disease vs platinum-resistant disease. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive liposome-encapsulated doxorubicin citrate IV over 60 minutes on day 1 and gemcitabine hydrochloride IV over 30 minutes on days 1 and 8. Treatment repeats every 3 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive liposome-encapsulated doxorubicin citrate IV over 60 minutes on day 1. Treatment repeats every 3 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.

Patients who experience clinical benefit after completion of 6 courses of chemotherapy may continue therapy at the discretion of the investigator.

Patients complete quality-of-life questionnaires (EORTC-QLQ30 and QLQ-OV28) at baseline, during, and after completion of study therapy. After completion of study treatment, patients are followed up every 3 months for up to 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ovarian epithelial, fallopian tube, or primary peritoneal cavity cancer
* Progression or recurrence during first-line platinum-based chemotherapy (platinum-refractory disease) OR progression or recurrence during the first 6 months following the end of the last platinum-containing chemotherapy (platinum-resistant disease)
* Meets ≥ 1 of the following criteria:

  * Measurable metastatic disease on CT or MRI scan, ultrasound, or chest x-ray
  * Evaluable disease on CT/MRI scan (e.g., ascites or pleural effusion) or chest x-ray (e.g., pleural effusion)
  * Tumor marker progression (CA-125) according to Rustin criteria, meeting 1 of the following criteria:

    * CA-125 > 2 times upper limit of normal (UNL)
    * CA-125 > 2 times nadir value on two occasions
* No ovarian carcinosarcoma (malignant mixed Müllerian tumor) or pure sarcoma

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* Life expectancy ≥ 3 months
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 10 g/dL
* Neutrophil count ≥ 1.5 x 10³/mm³
* Serum creatinine < 1.5 times ULN
* Bilirubin < 1.5 times ULN (< 2.5 times ULN if liver metastases are present)
* AST/ALT < 2.5 times ULN (unless caused by parenchymal liver metastases)
* No childbearing capacity
* LVEF ≥ 50% by ECHO or MUGA scan
* No significant comorbidity (e.g., uncontrolled infection, clinical signs of cardiac insufficiency, history of myocardial infarction, or cardiac rhythmic disorders [NYHA class III-IV disease])
* No known hypersensitivity to study drugs
* No active secondary malignant tumor within the past 5 years (e.g., metastases from primary breast cancer)
* No condition (medical, social, or psychological), that would prevent adequate follow-up

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy with pegylated liposomal doxorubicin hydrochloride, other anthracyclines, or gemcitabine hydrochloride
* No other concurrent tumor-specific therapy for ovarian cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2009-07; Primary Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Remission rates (complete response and partial response)

SECONDARY OUTCOMES:
Quality of life as measured by EORTC-QLQ30 and QLQ-OV28 questionnaires
Progression-free survival
Overall survival
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Alain Zeimet, Principal Investigator — Medical University Innsbruck
Locations (1):
- Innsbruck Universitaetsklinik, Innsbruck, Austria